CLINICAL TRIAL: NCT04126642
Title: Project Persist: mHealth for Cancer Survivorship
Acronym: Persist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11273
Record Dates: First submitted 2019-09-18; First posted 2019-10-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Symptom Management; Reduce Treatment Non-adherence
Keywords: improve symptom management; reduce treatment non-adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assessment only group (Other): Standard care + Daily ecological momentary assessments (EMAs)
  Interventions: Behavioral: Assessment only group
- Intervention group (Experimental): Intervention group will receive same measures and interventions as the assessment only group AND will receive messaging that is tailored to patient responses on EMAs. When participants provide a pattern of responses that are suggestive of heightened emotional distress, they will receive feedback and/or a prompt to complete one of the self-management exercise. The app will prompt participants to complete a brief educational video on relaxation strategies and guided relaxation exercises. Participants will have access to: 1) a "Help me Cope" button in the app that contains links to evidenced-based self-management techniques, and 2) a "Contact Counselor" button that will send a secure email to a study psychologist requesting a call. Participants will receive a coping focused message at the completion of the "Report Distress" EMAs. Participants can access these on demand intervention components and review them at any time in addition to receiving the tailored intervention messages.
  Interventions: Behavioral: Intervention group

INTERVENTIONS:
Behavioral: Assessment only group — Individuals randomized to this group will receive radiation therapy as usual plus baseline, follow-up, and EMA assessments.
  Arms: Assessment only group
Behavioral: Intervention group — Individuals randomized to the intervention group will complete the same measures (in person and daily EMAs) as the assessment only group, but will additionally receive messaging that is tailored to patient responses on EMAs.
  Arms: Intervention group

SUMMARY:
Many studies have shown that anxiety and depression are associated with reduced treatment adherence and poor treatment outcomes among patients undergoing cancer treatments. Given the negative consequences of psychological symptoms for cancer patients, it is important to effectively identify and address emotional distress among cancer patients. However, many barriers exist that limit access to effective treatments. Mobile health (mHealth) technologies offer the potential for remote monitoring and on demand management of psychological needs among cancer patients. This pilot randomized controlled trial (RCT) will assess the initial feasibility of a phone-delivered intervention for anxiety and depressive symptoms among cancer patients that are receiving active radiation treatments. A total of 60 participants will be randomized to in-person and smartphone-based assessment only (n=30) or assessment plus smartphone-based intervention (n=30). Both groups will be followed for 8 weeks (6 weeks while undergoing radiation therapy for breast or gynecological cancer + 2 weeks following radiation therapy). It is expected that patients who are randomized to the intervention group will report that the smartphone app is easy to use, app content is useful, and will show greater improvements in reported anxiety, depression, and quality of life compared with the assessment only group. Data from this pilot study will be used to inform the development of mHealth interventions that will be tested in future fully powered RCTs.

DETAILED DESCRIPTION:
A total of 60 individuals will be recruited from the OU Medicine Radiation Oncology Clinic (radiation clinic). All participants will be adults who are beginning radiation treatments for breast, gynecological, and head and neck cancers. Eligible participants include adult males and females 18+ who are: 1) community dwelling, 2) diagnosed with a primary breast or gynecological or head and neck cancer, 3) ordered to receive radiation treatments during a minimum of 6 consecutive weeks, and 4) able to read at the 7th grade level, speak, and write English. Exclusion criteria include: 1) radiation treatment with primary palliative intent, 2) radiation treatment protocol occurring in a time period of less than 6 weeks, 3) severe visual impairment that limits mobile technology use (e.g, partial or full blindness), and 4) history of dementia or other major neurocognitive disorder. Potential participants will be referred to this study for screening from multiple sources including from radiation clinic staff and self-referral. Eligible participants will be identified by radiation oncologists and other radiation clinic staff during initial consult visit, who will alert study staff of potential participants. Flyers will also be used to advertise the study to potential study participants, who can discuss enrollment with radiation oncologists. Those interested in participating in this study will complete the informed consent process. Those who meet the study inclusion criteria will be randomized into the assessment only group (n=30) or the assessment + intervention group (n=30). All participants will complete a baseline assessment visit which includes completion of study questionnaires, downloading the study smartphone app onto personal or study provided smartphones, and training to complete the phone based surveys (EMAs). Consent, baseline assessment, and mobile health training will take place in a private or semi-private space in the radiation clinic and is estimated to take 60-90 minutes to complete. Radiation oncology providers will be blinded to patient group assignment, which will occur during the baseline visit. Participants will complete EMAs for 8 weeks. At the end of the 8-week data collection period, participants will complete a final study survey using the study smartphone application and participate in a telephone interview.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants include adults 18+ who are:

1. community dwelling
2. diagnosed with a primary breast or gynecological or head and neck cancer
3. ordered to receive radiation treatments during a minimum of 5-6 consecutive weeks
4. able to read at the 7th grade level, speak, and write English.
5. scheduled for 5-6 weeks of radiation therapy

Exclusion Criteria:

1. radiation treatment with primary palliative intent
2. radiation treatment protocol occurring in a time period of less than 6 weeks
3. severe visual impairment that limits mobile technology use (e.g, partial or full blindness)
4. history of dementia or other major neurocognitive disorder. There are no early termination criteria; however, individuals can elect to stop participation in mobile monitoring at any time.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Improvement of anxiety and depression in intervention group compared with the assessment only control group | 8 weeks
  The study plans to assess the differences between the 8 week and baseline values of scores from validated scales for evaluating anxiety (GAD7) and depression (PHQ and CESD). Exact 95% confidence intervals will be estimated for the difference between the 8 week and baseline scores in the intervention and control groups. The scale scores for anxiety and depression obtained from the EMA measurements will also be modeled, which are correlated within participants. Thus, we will use linear mixed model regression analysis (LMM) on these repeated measures, employing a random intercept or slope parameter, as appropriate, to examine changes in these measures over time in the two treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States